CLINICAL TRIAL: NCT03103685
Title: Effect of Continue vs. Stop P2Y12 Inhibitor on Bleeding in Patient Receiving Dual-antiplatelet Therapy Undergoing Dental Procedure.
Brief Title: Continue vs. Stop P2Y12 Inhibitor on Bleeding in Patient Receiving DAPT Undergoing Dental Procedure.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kultida Lertthanaphol, Cardiology Unit, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MED-2559-04408
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Dental Diseases; Antiplatelet Agents; Antiplatelet Drugs
Keywords: Dual antiplatelet therapy; Dental procedure
MeSH Terms: conditions — Stomatognathic Diseases | interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The dentist will be blind wheater the patient takes DAPT or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ASA alone (Placebo Comparator): The patient in this arm will be ask to stop P2Y12 inhibitor before dental procedure, 5 days for clopidogrel and ticagrelol and 7 days for prasugrel.
  Interventions: Drug: Clopidogrel
- Uninterrupted DAPT (Experimental): The patient in this arm will continue dual anti platelet until the date of dental procedure.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — The patient s in experimental arm will not be ask to stop P2Y12 inhibitor such as Clopidogrel, Prasugrel or Ticagrelor
  Other Names: Prasugrel; Ticagrelor

SUMMARY:
This is a prospective randomized open-label blinded endpoint (PROBE) The study will be conducted in Maharaj Nakorn Chiang Mai hospital. The patients with dual-antipletlet who need dental procedure between Febuary 2017 until Febuary 2018 will be included in the study. Baseline characteristics of the enrolled patients including bleeding complication will be collected in each patient. To compare rate of significant bleeding from dental procedure between patient who need two antiplatelet and who stop P2Y12 inhibitors before procedure.

DETAILED DESCRIPTION:
Treatment of coronary artery disease is re-open the occluded artery by many ways such as removed clot and coronary stenting. Which needed two antiplatelet after the procedure at least a month to a year. Some patient must have life long period to prevent the stent occlude and stenosis. But dental problem is commonly found in real life practice. Many people suffered from toothache and have to wait until a year, just to prevent bleeding. Physicians often be consulted with this dilemma. To continue there are some risk to bleed but discontinue antipletlet can cause recurrent myocardial ischemia. Which the highest risk factor of stent thrombosis is early stop anti platelet. Since there is no clinical practice guideline in Thailand, this study is to compare rate of dental bleeding between patient who continue two antoplatelet and who stop only P2Y12 inhibitor. The study include immediate bleeding, 24 hour and a week after procedure, follow up for major cardiovascular event such as myocardial ischemia, stroke and death. In order to create further clinical practice for this specific group.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Need DAPT
* Need to ybeperform dental procedure such as simple extraction, complex extraction, and also focal, multifocal and total gingival scaling

Exclusion Criteria:

* patient with coagulopathy
* patient with Hemophilia
* patient with cirrhosis and renal pailure( BUN > 60, Cr > 6.0)
* patient who unable to come for medical visit in emergency condition such as severe bleeding
* patient with severe disease eg. advance stage cancer.
* patient with history of ACS less than 6 month
* patient who was be PCI wit DESless than 6 month
* patient with DAPT but planned to be CABG within a year.
* patient with anticoagulant
* patient who've got bisphosphonate within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of prolong bleeding from dental procedure | immediate after 30 minute post procedure
  Observed bleeding at 30 minute after finish dental procedure for 30 minute.

SECONDARY OUTCOMES:
Incidence of severe bleeding | at more than 12 hour after dental procedure or large hepatoma, or ecchymosis, or bleeding that need ER visit.
  Observed severe bleeding at subacute to late phase after dental procedure.
Incidence of major adverse cardiovascular event (MACE) | 7 and 30 days after dental procedure, patient well be called, to check her/his status.
  montior MACE after stop P2Y12

CONTACTS AND LOCATIONS:
Overall Officials: Arintaya Phrommintikul, M.D., Study Director — Chiang Mai University

IPD SHARING:
Plan to Share IPD: No